CLINICAL TRIAL: NCT01421563
Title: A Randomized, Open-label, Two-Sequence, Two-Period Crossover Study to Assess the Pharmacokinetic Characteristics of Sarpogrelate HCl Controlled Release Tablet Compared With Sarpogrelate HCl Immediate Release Tablet in Healthy Male Subjects
Brief Title: Safety and Pharmacokinetic Characteristics of DP-R202 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DP-SACL-I-001
Record Dates: First submitted 2011-07-27; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anplag (Active Comparator)
  Interventions: Drug: Anplag
- DP-R202 (Experimental)
  Interventions: Drug: Anplag

INTERVENTIONS:
Drug: Anplag — Sarpogrelate HCl 300mg once a day or 100mg three times a day
  Other Names: DP-R202 : DP11002-2; Anplag : 0007

SUMMARY:
The purpose of this study is compare the safety and pharmacokinetic characteristics of DP-R202 (Sarpogrelate HCl 300mg, qd) with those of Anplag (Sarpogrelate HCl 100mg, tid) after oral administration in healthy male volunteers.

DETAILED DESCRIPTION:
The number of patient is thirthy-six.Patients were randomly assigned either anplag tablet(Sarpogrelate HCL 100mg, tid)first, DP-R202(Sarpogrelate HCL 300mg, qd) Second or DP-R202(Sarpogrelate HCL 300mg, qd) first, anplag tablet(Sarpogrelate HCL 100mg, tid) second.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of healthy volunteers

Exclusion Criteria:

* Hypersensitivity Reaction about Sarpogrelate HCL or other antiplatelets

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Cmax, AUClast | 24h

SECONDARY OUTCOMES:
tmax, t1/2, AUC0-∞ | 24h

CONTACTS AND LOCATIONS:
Overall Officials: JaeWook Ko, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea